CLINICAL TRIAL: NCT05638906
Title: Minimally Invasive Nasal Trabeculostomy - Performance and Safety Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanoculis Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMS EEU-4
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: This Study is Obtained Under Inclusion/ Exclusion Criteria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single-arm study with intra-subject comparisons (Experimental): Study eyes of subjects with uncontrolled (IOP > 20 mmHg) open-angle glaucoma (OAG), where IOP is not controlled when using maximum tolerated glaucoma medications.
  Interventions: Device: MINT

INTERVENTIONS:
Device: MINT — Mechanical rotation of the Surgical Device is achieved by the rotating system (i.e., Activation Device), which is comprised of: (1) Controller which dictates the activation pulse duration, the rotations per minute (RPM) and the forwards and backwards movement of the micro trephine; (2) Motor; and (3) Footswitch.

SUMMARY:
Minimally Invasive Nasal Trabeculostomy System is intended for the reduction of elevated Intraocular Pressure (IOP).

The system is a powered surgical device, designed to create trabeculostomy openings of ~100 microns diameter each, via an ab-interno approach, directly from the anterior chamber (AC) into Schlemm's canal (SC) by removing segments of the trabecular meshwork (TM) (i.e., an ab-interno nasal trabeculostomy). The ab-interno approach aims to decrease IOP by increasing aqueous outflow through a direct communication from the AC to the outer wall of SC and the collector channels.

The opening in the nasal TM to the SC is created by a sterile surgical instrument (the Surgical Device) made of stainless steel and plastic, which is coupled to a rotating system (the Activation Device). The Surgical Device of the Minimally Invasive Nasal Trabeculostomy System consists of a stainless steel micro trephine, covered by a small needle-shaped sleeve with a rotating mechanism behind it. While being rotated, the Surgical Device enters and moves along the TM, removing TM tissue with minimal collateral damage.

Mechanical rotation of the Surgical Device is achieved by the rotating system (i.e., Activation Device), which is comprised of: (1) Controller which dictates the activation pulse duration, the rotations per minute (RPM) and the forwards and backwards movement of the micro trephine; (2) Motor; and (3) Footswitch.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female ≥ 18 years to ≤ 85 years old 2. Unsatisfactory IOP level, i.e., IOP ≥21 mmHg, at the screening visit in the study eye 3. Manifest open angle glaucoma (OAG) with typical disc or visual field changes and open iridocorneal angle in the study eye (in accordance with European Glaucoma Society (EGS) criteria 1) 4. Optic nerve appearance characteristic of glaucoma in the study eye 5. Shaffer grade ≥ III in all four angle quadrants in the study eye 6. Subject is treated with 0 to 5 hypotensive medications in the study eye 7. Subject is able and willing to attend all scheduled follow-up exams 8. Subject understands and signs the informed consent

Exclusion Criteria:

* 1. Ocular conditions with a poorer prognosis in the fellow eye than in the study eye 2. Closed angle forms of glaucoma in either eye unless scheduled for cataract surgery immediately prior to the Minimally Invasive Nasal Trabeculostomy procedure or the study eye is pseudophakic with posterior chamber intraocular lens (PCIOL) 3. Congenital or developmental glaucoma in either eye 4. Fixation threatening visual-field defects or IOP ≥40 mmHg in the study eye

  1. Other secondary glaucoma (such as neovascular, uveitic, lens-induced, trauma-induced, or glaucoma associated with increased episcleral venous pressure) in the study eye
  2. Peripheral anterior synechiae (PAS), rubeosis or other angle abnormalities in the study eye
  3. Subject has history of penetrating keratoplasty (PKP)
  4. Any previous surgery in the study eye (at the access site of the Minimally Invasive Nasal Trabeculostomy System application), where the conjunctiva is not intact and elastic (except for clear corneal cataract surgery)
  5. Any ocular disease or history in study eye such as severe dry eye, active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, and ocular pathology that may interfere with accurate IOP measurements
  6. Prior surgery for an ab-interno or ab-externo device implanted in or through the Schlemm's canal in the study eye.
  7. Best-corrected visual acuity worse than 20/40 (Snellen equivalent) in the fellow eye
  8. History of idiopathic or autoimmune uveitis in either eye
  9. Severe trauma in study eye
  10. Active iris neovascularization, previous cyclodestructive procedure, prior scleral buckling procedure, presence of silicone oil, need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery in study eye within 12 month period
  11. Vitreous present in anterior chamber, prior vitrectomy or vitreous hemorrhage in study eye
  12. Aphakia
  13. Prior vitreoretinal surgery in study eye
  14. Clinically significant ocular inflammation or infection within 90 days prior to screening
  15. Unable to discontinue use of blood thinners in accordance with surgeon's standard preoperative instructions
  16. Uncontrolled systemic disease that in the opinion of the investigator would put the subject's health at risk and/or prevent the subject from completing all study visits
  17. Current participation or participation in another investigational drug or device clinical trial within the last 30 days before screening visit
  18. Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieved a 20% or greater reduction in IOP from Baseline on the same or fewer number of medications [time frame: 24 weeks | 24 months
  • Proportion of subjects achieving a 20% or greater reduction in IOP from baseline on the same or fewer number of medications. Subjects who will undergo a glaucoma-related secondary surgical intervention prior to the 24 weeks visit will be considered failures in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- S.V.Malayan'S Eye Center, Yerevan, Armenia

REFERENCES:
- [Derived] Voskanyan L, Miroyan H, Papoyan V, Babayan H, Grover DS. Performance and Safety of Minimally Invasive Nasal Trabeculostomy (MINT) in Open-Angle Glaucoma: A 12-month Open-Label Study on Patients with No Other Glaucoma Surgeries. Clin Ophthalmol. 2025 Dec 19;19:4841-4853. doi: 10.2147/OPTH.S538801. eCollection 2025. PMID 41446893